CLINICAL TRIAL: NCT04415905
Title: Comparison of Optic Nerve Sheath Diameter in Children Receiving Caudal Block According to Anesthetic Agents: Total Intravenous Anesthesia vs. Volatile Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4-2020-0061
Record Dates: First submitted 2020-05-28; First posted 2020-06-04 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Caudal Block for Postoperative Analgesia
Keywords: Caudal block; Intracranial pressure; Propofol; Sevoflurane; Ultrasound
MeSH Terms: interventions — Propofol; Sevoflurane

STUDY DESIGN:
Intervention Model Description: There are 2 groups according to the type of main anesthetic agent. P group are anesthetized with propofol, so are S group with sevoflurane.
Who Masked: Outcomes Assessor
Masking Description: Anesthesia machine and infusion pumps are shielded from assessors who measure ONSD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group P (Experimental): The participants in the group P are anesthetized with propofol.
  Interventions: Drug: Propofol
- group S (Active Comparator): The participants in the group S are anesthetized with sevoflurane.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — The participants in the group P are anesthetized with propofol
  Arms: group P
Drug: Sevoflurane — The participants in the group S are anesthetized with sevoflurane.
  Arms: group S

SUMMARY:
Caudal block is commonly used for postoperative analgesia in paediatric patients. A higher volume (1.5 ml/kg) of local anaesthetic for caudal block has been reported to not only increase the level of cranial spread but also provide better quality and longer duration of analgesia in comparison with the conventional volume (1.0 ml/kg). However, caudal block with a high volume of local anaesthetic can increase intracranial pressure (ICP). Previous studies have shown that propofol anesthesia lowers ICP when compared with volatile anesthesia. Therefore, this study was designed to test if propofol can reduce the magnitude of ICP increase following caudal block when compared with a volatile anesthetic, sevoflurane. There is increasing evidence that optic nerve sheath diameter (ONSD) measured by ultrasonography correlates with degree of ICP and is able to detect intracranial hypertension. Therefore, ONSD will be measured as a surrogate of ICP.

DETAILED DESCRIPTION:
Equal number of patients are randomly assigned to the P or S group. The participants in the P and S group are anesthetized with propofol and sevoflurane, respectively. Irrespective of assigned group, all participants receive caudal block with 1.5 ml/kg of 0.15% ropivacaine (up to 30 ml per individual participant). All anesthetic procedures except for main anesthetic agent are the same in all participants. ONSD is measured at the following time points: before (T0), immediately after (T1), and 10 min (T2) and 30 min(T3) after caudal block. Two measurements of each optic nerve sheath are acquired in each eye. The mean value of the four measurements is considered as the ONSD at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Among children undergoing urological surgery, patients, 36 to 72-months-old
* Body weight less than 20 kg (The limit on body weight is set because the maximum volume of local anaesthetic for caudal block in children is restricted to 30 ml.)
* Treatment plan for caudal block for analgesia, are enrolled.

Exclusion Criteria:

* Symptoms or signs of spinal anomalies or infection at the sacral region
* Coagulopathy
* Increased ICP
* Ophthalmic diseases
* History of increased ICP

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-03-02 (Actual)

PRIMARY OUTCOMES:
ONSD | before (T0) caudal block.
  ONSD is a surrogate for ICP. ONSD was measured by transorbital sonography. Transorbital sonography is performed using a linear 6-13 Hz probe. After applying a thick layer of sterile coupling gel on the closed upper eyelid, the probe is placed gently without exerting pressure. Axial images of the orbit are acquired in the plane of the optic nerve, and ONSD is measured 3mm posterior to the optic nerve head as described previously.
ONSD | immediately after (T1) caudal block.
  ONSD is a surrogate for ICP. ONSD was measured by transorbital sonography. Transorbital sonography is performed using a linear 6-13 Hz probe. After applying a thick layer of sterile coupling gel on the closed upper eyelid, the probe is placed gently without exerting pressure. Axial images of the orbit are acquired in the plane of the optic nerve, and ONSD is measured 3mm posterior to the optic nerve head as described previously.
ONSD | 10 minutes (T2) after caudal block.
  ONSD is a surrogate for ICP. ONSD was measured by transorbital sonography. Transorbital sonography is performed using a linear 6-13 Hz probe. After applying a thick layer of sterile coupling gel on the closed upper eyelid, the probe is placed gently without exerting pressure. Axial images of the orbit are acquired in the plane of the optic nerve, and ONSD is measured 3mm posterior to the optic nerve head as described previously.
ONSD | 30 minutes (T3) after caudal block.
  ONSD is a surrogate for ICP. ONSD was measured by transorbital sonography. Transorbital sonography is performed using a linear 6-13 Hz probe. After applying a thick layer of sterile coupling gel on the closed upper eyelid, the probe is placed gently without exerting pressure. Axial images of the orbit are acquired in the plane of the optic nerve, and ONSD is measured 3mm posterior to the optic nerve head as described previously.

SECONDARY OUTCOMES:
The variables affecting ICP : Heart rate (beats per minute) | before (T0) caudal block.
The variables affecting ICP : Heart rate (beats per minute) | immediately after (T1) caudal block.
The variables affecting ICP : Heart rate (beats per minute) | 10 minutes (T2) after caudal block.
The variables affecting ICP : Heart rate (beats per minute) | 30 minutes (T3) after caudal block.
The variables affecting ICP : Mean arterial pressure (mmHg) | before (T0) caudal block.
The variables affecting ICP : Mean arterial pressure (mmHg) | immediately after (T1) caudal block.
The variables affecting ICP : Mean arterial pressure (mmHg) | 10 minutes (T2) after caudal block.
The variables affecting ICP : Mean arterial pressure (mmHg) | 30 minutes (T3) after caudal block.
The variables affecting ICP : End-tidal carbon dioxide partial pressure (mmHg) | before (T0) caudal block.
The variables affecting ICP : End-tidal carbon dioxide partial pressure (mmHg) | immediately after (T1) caudal block.
The variables affecting ICP : End-tidal carbon dioxide partial pressure (mmHg) | 10 minutes (T2) after caudal block.
The variables affecting ICP : End-tidal carbon dioxide partial pressure (mmHg) | 30 minutes (T3) after caudal block.
The variables affecting ICP : End-tidal sevoflurane concentration (volume %) | before (T0) caudal block.
The variables affecting ICP : End-tidal sevoflurane concentration (volume %) | immediately after (T1) caudal block.
The variables affecting ICP : End-tidal sevoflurane concentration (volume %) | 10 minutes (T2) after caudal block.
The variables affecting ICP : End-tidal sevoflurane concentration (volume %) | 30 minutes (T3) after caudal block.
The variables affecting ICP : Estimated propofol effect-site concentration (μg/ml) | before (T0) caudal block.
The variables affecting ICP : Estimated propofol effect-site concentration (μg/ml) | immediately after (T1) caudal block.
The variables affecting ICP : Estimated propofol effect-site concentration (μg/ml) | 10 minutes (T2) after caudal block.
The variables affecting ICP : Estimated propofol effect-site concentration (μg/ml) | 30 minutes (T3) after caudal block.
The variables affecting ICP : Body temperature (℃) | before (T0) caudal block.
The variables affecting ICP : Body temperature (℃) | immediately after (T1) caudal block.
The variables affecting ICP : Body temperature (℃) | 10 minutes (T2) after caudal block.
The variables affecting ICP : Body temperature (℃) | 30 minutes (T3) after caudal block.
The variables affecting ICP : Peak inspiratory pressure (mmHg) | before (T0) caudal block.
The variables affecting ICP : Peak inspiratory pressure (mmHg) | immediately after (T1) caudal block.
The variables affecting ICP : Peak inspiratory pressure (mmHg) | 10 minutes (T2) after caudal block.
The variables affecting ICP : Peak inspiratory pressure (mmHg) | 30 minutes (T3) after caudal block.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No